CLINICAL TRIAL: NCT06022549
Title: Effects of mHealth Message on Metabolic Syndrome and Bone Loss of HIV Infected Persons in Taiwan
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University (Other)
Responsible Party: Principal Investigator, Piao-Yi Chiou, Associate Professor, National Taiwan University
Other Study IDs: 202301HM003
Record Dates: First submitted 2023-08-25; First posted 2023-09-05 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Hiv
Keywords: HIV-infected persons; Metabolic syndrome
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With improved AIDS treatment leading to extended survival, HIV-infected individuals face a higher metabolic syndrome incidence. This study aims to determine the prevalence of Non-AIDS related Comorbidities (NARC) in HIV-infected individuals. Using purposive and snowball sampling, the cross-sectional survey targets 400 HIV-infected individuals aged 30 and above. Data collection includes demographics, physical activity, nutrition, depression, and physiological measurements. Analyzing the data through statistical tests and structural equation modeling, the study aims to provide precise care recommendations for preventive medicine and healthy aging in this population.

DETAILED DESCRIPTION:
With the success of treatment, the survival period of Acquired immunodeficiency syndrome (AIDS) patients is prolonged. Compared with non-HIV-infected persons of the same age, HIV-infected persons have a relatively higher incidence of metabolic syndrome (MS). The main purpose of this study is to estimate the prevalence of common Non-AIDS related Comorbidities (NARC) among HIV-infected persons This study is a cross-sectional survey, purposive and snowball sampling will be applied. The recruitment information is released through channels such as AIDS case managers, AIDS non-government organizations, and social networks of HIV-infected people all around Taiwan. The expected sample size is 400 HIV-infected persons over the age of 30, after signing a written consent form, a test will be conducted, including the collection of demographic data, questionnaire data collection with physical activity scale, mini-nutrition assessment scale, and depression self-test scale, and measurement of physiological parameters using instruments including a gripper, body composition meter, sphygmomanometer, blood glucose, and lipid monitor, tape measure. The Chi-square test and independent sample T-test are used to compare the differences in the categorical and continuous data of each variable, and the structural equation model is used to conduct path analysis of the research framework. The research results can be used as precise care recommendations for the development of preventive medicine and healthy aging for HIV-infected persons.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected persons over the age of 30

Exclusion Criteria:

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected persons over the age of 30
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Mini Nutritional Assessment | 1 year
  The points of this assessment is from 0 to 30. The points over 23.5 mean normal nutritional status, 17~23.5 points mean at risk of malnutrition, less 7 points mean malnourished.
International Physical Activity Questionnaire | 1 year
  It is a self-administered survey used to assess an individual's physical activity levels. It aims to measure the amount of physical activity a person engages in across various domains of life, including work, transportation, household chores, and leisure time.
  The IPAQ typically asks participants about the duration and frequency of their physical activities in the past seven days. The MET-minutes per week score is calculated by multiplying the minutes spent in each activity intensity level by the MET value associated with that activity and then summing these values across all activities.
  The interpretation of MET-minutes per week is as follows:
  Low activity: Below 600 MET-minutes per week Moderate activity: 600 to 3000 MET-minutes per week High activity: More than 3000 MET-minutes per week
Patient Health Questionnaire-9 | 1 year
  The Patient Health Questionnaire-9 (PHQ-9) is a self-report assessment tool commonly used to screen and measure the severity of depression symptoms in individuals. It consists of 9 items or questions, each assessing different aspects of depression such as mood, energy level, and concentration.
  The PHQ-9 scores each item on a scale from 0 (not at all) to 3 (nearly every day), with a maximum total score of 27. Higher scores on the PHQ-9 indicate more severe depressive symptoms, while lower scores suggest milder or no depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: PIAO-YI CHIOU, doctoral, Study Director — National Taiwan University, College of Medicine, School of Nursing
Locations (1):
- National Taiwan University, College of Medicine, School of Nursing, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided